CLINICAL TRIAL: NCT03938519
Title: Attitude of Dentists Towards Radiography, Radiographic Equipment, Radiation Protection and Choice of Digital Imaging Methods in Cairo, Egypt-A Questionnaire Based Cross-Sectional Study
Brief Title: Attitude of Dentists About Radiography, Radiographic Equipment and Radiation Protection in Egypt
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hazem Elsaeed Fouda, Master degree student, Cairo University
Other Study IDs: ORAD 7-2-1
Record Dates: First submitted 2019-04-26; First posted 2019-05-06 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Limited Information on Dental Radiography in Egypt
Keywords: survey; questionnaire; radiation protection; dental

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A Survey for Attitude and Awareness about radiography, radiographic equipment and radiation protection among dentists in Egypt

DETAILED DESCRIPTION:
Settings:

* The sample size has been calculated according to population of dentists recorded in the Egyptian Dental Syndicate.
* Keeping in mind the difficulty in obtaining registered dentists' names and postal addresses, unreliable postal system and anticipated low response rate to a postal survey, it was decided to deliver and collect the questionnaires by hand.
* To prepare the questionnaire, a review of the literature was performed and the variables were determined.
* Questionnaires have been created in two forms according to the Type of Image receptor
* Form A will be for Dentists who use Film Packets
* Form B will be for Dentists who use Digital receptors
* The questionnaire includes a covering letter with an informed consent
* The cover letter provided in both English and Arabic, explaining the MSc research project and details of the project supervisor. The cover letter stated that by completing the questionnaire the participating dentists would be giving their voluntary consent to participate in the study.

Data Sources / Measurements:

* Some of the questions will be answered with either yes, no or an open alternative. For some of the questions several answers will be given; others were designed as an array of claims using a rating scale
* Questionnaires will be distributed randomly and manually on multiple refresher courses and congresses throughout the country.
* If necessary by a personal interview. The interview involved the author asking the dentists questions directly and noting down the replies without any elaboration or further explanation of the questionnaire.
* Forms of Questionnaires will be distributed according to dentist's choice in the first question which will be asked orally about the type of receptor is used during routine practice
* Paper based questionnaire will be distributed in envelope and returned to the researcher closed non marked to ensure confidentiality
* Prospective Data Analysis will be performed after the Questionnaires being collected
* The study will be conducted in department of Oral and Maxillofacial Radiology, Faculty of Dentistry, Cairo University.
* The guidelines were derived from the American Dental Association 2006 recommendations

Addressing potential sources of bias

* Bias of selection: Questionnaires will be distributed randomly and manually on multiple refresher courses and congresses throughout the country.
* Bias of Performance: Paper based questionnaire will be distributed in envelope and returned to the researcher closed non marked

ELIGIBILITY:
Dentists for assessment of attitude towards Oral Radiology will be selected according to the following criteria:

Inclusion criteria:

* All graduated dentists without limit in degree and qualifications
* Males and Females
* Dentists registered in Egyptian Dental Syndicate
* Dentists work in Private dental clinics
* Dentists work in Governmental sector
* Intern students

Exclusion criteria:

* Undergraduate students
* Individuals are not interested in the study

Ages: 24 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dentists Work in Egypt
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Knowledge and attitude towards Dental Radiology | up to 2020
  A survey questionnaire on the following criteria
  * Primary knowledge about the radiation protection
  * Selection criteria
  * Radiographic equipment and techniques
  * Method of patient and personnel protection
  * Management of radiographic waste. Dentists will have to answer on multiple choices questions
  Measuring Unit:
  Categorical nominal data (A rating scale for awareness ) High, Moderate and Low

SECONDARY OUTCOMES:
Practice and opinions about Digital Radiography | up to 2020
  A survey questionnaire on the following criteria :
  * percentage of dentists had made the transition to digital radiography
  * the type of detector used
  * problems experienced with digital radiography,
  * reasons for choosing digital technology
  * reasons for not choosing digital technique Some of the questions could be answered with either yes, no or an open alternative. For some of the questions several answers could be given
  Measuring Unit:
  Categorical nominal data (%)